CLINICAL TRIAL: NCT02671955
Title: An Open-label, First-in-Human, Phase 1 Study of the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-61610588, a Fully Human IgG1 Kappa Anti-VISTA (V-domain Ig Suppressor of T-cell Activation) Monoclonal Antibody, in Subjects With Advanced Cancer
Brief Title: A Study of Safety, Pharmacokinetics, Pharmacodynamics of JNJ-61610588 in Participants With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Janssen business decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108083; 61610588LUC1001 (Other: Janssen Research & Development, LLC); 2016-001903-22 (EudraCT Number)
Record Dates: First submitted 2016-01-11; First posted 2016-02-02 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; JNJ-61610588

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (Experimental): Participants with advanced solid tumors will receive intravenous infusions of JNJ-61610588 until disease progression. Dose escalation will continue until the maximum tolerated dose is reached.
  Interventions: Drug: JNJ-61610588
- Part 2: Biomarker Evaluation (Experimental): Participants with metastatic Non-small Cell Lung Cancer (NSCLC) will receive intravenous infusion of JNJ-61610588 at or below the recommended Phase 2 dose (RP2D) until disease progression.
  Interventions: Drug: JNJ-61610588
- Part 3: Dose Expansion (Experimental): Participants with metastatic Non-small Cell Lung Cancer (NSCLC) will receive intravenous infusion of JNJ-61610588 at the recommended Phase 2 dose (RP2D) until disease progression.
  Interventions: Drug: JNJ-61610588
- Part 4: Dose Expansion (Experimental): Participants with advanced solid tumors will receive intravenous infusion of JNJ-61610588 at the recommended Phase 2 dose (RP2D) until disease progression.
  Interventions: Drug: JNJ-61610588

INTERVENTIONS:
Drug: JNJ-61610588 — Participants will receive intravenous infusions of JNJ-61610588 until disease progression.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of JNJ-61610588 in participants with advanced cancer in order to determine a recommended Phase 2 dose (RP2D) for further evaluation in specific tumor types.

DETAILED DESCRIPTION:
The purpose of this study is to see if JNJ-61610588 is safe and useful for treating participants with advanced cancer. This study consists of up to 4 parts. Part 1 will determine what dose of JNJ-61610588 can be given safely to advanced cancer participants. Part 2 will look at how participants with metastatic non-small cell lung cancer respond to a safe dose of JNJ-61610588. Parts 3 and 4 will test whether the dose of JNJ-61610588 identified in Part 1 is a safe and effective therapy for participants with specific types of advanced cancers (lung, pancreas, cervical, colorectal, head and neck). Participants will receive study drug in an outpatient setting. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a solid tumor. Parts 2 and 3 are limited to participants with non-small cell lung cancer. Part 4 is limited to participants with small cell lung, head and neck, pancreatic, colorectal, and cervical cancers
* Tumor progression following at least one prior standard therapy
* The participant has a radiographically measurable tumor. Evaluable disease is acceptable for Part 1 only
* The participant is willing to consent to provide a tumor tissue sample (fresh biopsy) before (Parts 2 and 3) and after (Part 2 only) receiving the study drug
* The participant is able to carry out daily life activities without difficulty
* The participant does not have significant side effects from previous anti-cancer treatment
* The participant has adequate organ and blood cell counts
* Sexually active participants must use medically acceptable methods of contraception during the course of this study

Exclusion Criteria:

* The participant has a history of major surgery or treatment other cancer therapy within 2-6 weeks before starting the study
* The participant has an untreated brain tumor
* Current severe, uncontrolled systemic disease including an ongoing, active infection requiring treatment with antibiotics
* The participant has high blood pressure or diabetes that is not well-controlled with medication
* History of clinically significant heart problems
* History of severe side effects toimmunotherapy
* The participant is pregnant, breastfeeding, or planning to become pregnant or father a child
* Positive for Hepatitis B, Hepatitis C, or HIV
* The participant has received anticoagulant therapy with the exception of aspirin within 1 week of starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Frequency of Dose Limiting Toxicity (DLT) | Approximately 2.5 years
  The Dose Limiting Toxicity (DLT) is based on adverse events and includes unacceptable hematologic toxicity, unacceptable non-hematologic toxicity of Grade 3 or higher, and treatment delay greater than 2 weeks.
Number of Participants with Adverse Events (AEs) and Serious AEs | Approximately 2.5 years
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Change From Baseline in Pharmacodynamic Blood Biomarkers- Total Blood Cell Counts | Approximately 2.5 years
  Standard hematology laboratory tests will be used to evaluate total blood cell counts in blood samples collected pre- and posttreatment.
Change From Baseline in Pharmacodynamic Blood Biomarkers- Markers of Monocyte Activation | Approximately 2.5 years
  Flow cytometry will be used to evaluate markers of monocyte activation in blood samples collected pre- and posttreatment.
Change From Baseline in Pharmacodynamic Blood Biomarkers- Markers of T Cell Activation | Approximately 2.5 years
  Flow cytometry will be used to evaluate markers of T cell activation in blood samples collected pre- and posttreatment.
Change From Baseline in Pharmacodynamic Tissue Biomarkers- Protein Expression of VISTA (V-domain Ig suppressor of T cell activation) | Approximately 2.5 years
  Pre- and posttreatment tissue samples will be stained by immunohistochemistry for protein expression of VISTA.
Change From Baseline in Pharmacodynamic Tissue Biomarkers- Markers Associated With Immune Infiltrate Including CD3, CD4, CD8, Forkhead box P3, CD68, and PD-L1. | Approximately 2.5 years
  Pre- and posttreatment tissue samples will be stained by immunohistochemistry for markers associated with immune infiltrate including CD3, CD4, CD8, forkhead box P3, CD68, and PD-L1.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of JNJ-61610588 | Approximately 2.5 years
  The Cmax is the maximum observed serum concentration of JNJ-61610588.
Elimination Half-Life (t1/2) | Approximately 2.5 years
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Area Under the Serum Concentration-Time Curve From t1 to t2 Time (AUC[t1-t2]) of JNJ-61610588 | Approximately 2.5 years
  The AUC(t1-t2) is the area under the serum JNJ-61610588 concentration-time curve from time t1 to t2.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Approximately 2.5 years
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Number of Participants With Anti-JNJ-61610588 Antibodies | Approximately 2.5 years
  Plasma levels of antibodies to JNJ-61610588 for evaluation of potential immunogenicity.
Assessment of Anti-Tumor Activity, as Assessed by the Overall Response Rate (ORR) | Approximately 2.5 years
  Anti-tumour activity as assessed by the ORR based on Response Evaluation Criteria in Solid Tumours (RECIST), version 1.1.
Assessment of Anti-Tumor Activity, as Assessed by the Overall Response Rate (ORR) | Approximately 2.5 years
  Anti-tumour activity as assessed by the ORR based on Immune-Related Response Criteria (irRC).
Assessment of Anti-Tumor Activity, as Assessed by Duration of Response | Approximately 2.5 years
  Anti-tumour activity as assessed by the duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - New York, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas